CLINICAL TRIAL: NCT02026089
Title: Persistence of Varicella Immunity in Hospital Employees Receiving Varicella Vaccine
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Unforeseen reduction of recruitment resource.
Sponsor: University of Colorado, Denver (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 13-1380
Record Dates: First submitted 2013-12-23; First posted 2014-01-01 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Persistence of Varicella Immunity
MeSH Terms: interventions — Chickenpox Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sero-positive for varicella at least 5 years prior (No Intervention): No treatment
- Varicella vaccine (Active Comparator): One dose varicella vaccine (Varivax).
  Interventions: Biological: Varicella vaccine

INTERVENTIONS:
Biological: Varicella vaccine — Varivax 0.5ml subcutaneous injection
  Other Names: Varivax
  Arms: Varicella vaccine

SUMMARY:
The purpose of the study is to learn more abou how the immune system responds to the chickenpox vaccine in adults who had never had chickenpox as a child and were then vaccinated as an adult. The study aims to learn more about the strength and duration of the protection provided by the vaccine in adults, and to observe the immune response to an additional dose of chickenpox vaccine in adults who had received the vaccine at least 5 years earlier. This is especially relevant to workers in a hospital who may be exposed to chickenpox.

DETAILED DESCRIPTION:
The population will be employees who were previously evaluated in the pre-employment phase by the Occupational Health Clinic (OHC) of Colorado Children's Hospital (CHC) from 2004 until 2009 and were found to be seronegative for varicella antibody at that time and were thus vaccinated per CHC protocol. Additionally, a matching number of comparator subjects who were positive for varicella antibody at the pre-employment phase will be selected from the same pool (2004-2009).

Subject participation will last up to 6 months. Subjects will be enrolled into one of two study groups:

* Group 1 consisting of 50 subjects who tested seronegative for varicella antibody and received varicella vaccine to meet employment criteria at least 5 years previously; and
* Group 2 consisting of 50 subjects who had natural varicella infection and thus tested seropositive for varicella antibody at least 5 years previously.

Group 1 subjects will receive 1 additional dose (lifetime total will be 2 or 3) of varicella vaccine (Varivax) and participate in a total of 4 study visits over a period of 6 months. Before receiving the dose of varicella vaccine at Day 1, Group 1 subjects will be given the CDC Vaccine Information Sheet for varicella vaccine. Study staff will review this with the subject to assure understanding prior to administering vaccine. Vaccination will occur after eligibility criteria have been confirmed and completion of a urine pregnancy test -with a negative result - on females of childbearing potential. Following administration of the varicella vaccine, the subject will be observed in the clinic for at least 15 minutes for safety. Blood (60 ml per sample) will be collected from all Group 1 subjects on Day 1 immediately prior to vaccination, and at Day 7(±2), Day 30(±7) and Day 180(±14) in order to measure VZV-specific antibody, antibody avidity, and cell-mediated immunity by the methods indicated above. Subjects receiving a third lifetime dose of Varivax will be asked to complete a diary for 5 days after vaccination to track anticipated and unanticipated reactions to the vaccine.

Group 2 subjects, the comparator group, will receive no vaccine and will only participate in the first visit for a blood draw. Blood (60 ml) will be collected from Group 2 participants only at Day 1. Subject information to be recorded includes age; gender; varicella vaccine history at the OHC; age vaccinated (calculate interval since vaccination); the number of doses (1 vs 2) received; and any exposure to varicella or HZ (including involvement in any CHC outbreak work-up).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Group 1: * Evaluated in Occupational Health Clinic (OHC) for employment from 2004-2009 and found to be seronegative for varicella.

  * Received at least one varicella vaccination to meet employment criteria at least 5 year prior to enrollment.
  * Subject is afebrile (<100.4F oral) on day of vaccination.
* Group 2: * Evaluated in OHC for employment from 2004 -2009 and found to be seropositive for varicella.

Exclusion Criteria:

* Immune suppressed or receiving immune suppressive treatment
* Pregnant, breastfeeding or plan to become pregnant within 6 weeks after receiving varicella vaccine.
* Receiving antiviral medications active against varicella virus within 3 days before varicella vaccination until 10 days after varicella vaccination.
* Receipt of any vaccine within 2 weeks before enrollment or expected receipt within 6 weeks after vaccination.
* Receipt of any immunoglobulins or blood products within 5 months prior to study enrollment or expected receipt prior to last visit.
* History of hypersensitivity reaction to any vaccine component (including gelatin), or an anaphylactic/anaphylactoid reaction to neomycin.
* History of chickenpox or shingles since pre-employment serology testing.
* Receipt of any additional varicella or zoster vaccine since vaccination under hospital policy and procedure guidelines.
* Currently participating in any other studies with an investigational compound within 30 days of signing the consent and throughout participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Determine the proportion of employees who 5 years previously received varicella vaccine at the time of employment who no longer have varicella-specific antibody. | Outcome measure data obtained at visit 1; assessed in the aggregate 3-6 months after completion of study.
  VZV-specific antibody measured by a sensitive gp-ELISA method at CDC

SECONDARY OUTCOMES:
Determine the avidity (strength with which the vaccine induced antibody binds to the varicella antigen) of varicella-specific antibody in vaccinated employees. | Outcome measure data obtained at visit 1; assessed in the aggregate 3-6 months after completion of study.
  Avidity in these employees will be compared to the avidity of antibody in employees who did hot require vaccination because of natural immunity.

OTHER OUTCOMES:
Determine the varicella-specific T-cell and B-cell responses in vaccinees. | At 7 and 30 days post-vaccination
  Responses will be compared to those present in employees who did not require vaccination because of natural immunity.

CONTACTS AND LOCATIONS:
Overall Officials: Myron J Levin, MD, Principal Investigator — University of Colorado School of Medicine
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No